CLINICAL TRIAL: NCT04238195
Title: A Single-Dose, Randomized, Placebo- and Active-Control, Four-Way, Cross-Over Study for the Evaluation of the Effect of Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) on the QT/QTc Intervals in Adult Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Spero Therapeutics (Industry)
Collaborators: Celerion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: SPR994-104
Record Dates: First submitted 2020-01-16; First posted 2020-01-23 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: TQT Study
Keywords: TQT
MeSH Terms: interventions — tebipenem; Moxifloxacin

STUDY DESIGN:
Intervention Model Description: Over 4 separate treatment periods, each separated by a 7-day washout period, all subjects will receive a single dose of 4 different study treatments.The design is constructed from three 4x4 Latin Squares balanced for carry-over effects.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A computerized randomization scheme will be created by a CRO-statistician and it shall be considered blinded (as per the following).
  The randomization is available only to the pharmacy staff that is preparing the drug who will not be involved in any other aspect of the study including administration of the drug. The randomization will also be available to the bioanalytical laboratory as sample analyses will be treatment-dependent. It will not be made available to the Sponsor, subjects, or members of the staff responsible for the monitoring and evaluation of safety assessments.
  On Day 1 of each period, subjects will receive a single oral therapeutic dose of TBPM-PI-HBr (Treatment A), supratherapeutic dose of TBPM-PI-HBr (Treatment B), placebo (Treatment C), or moxifloxacin (Treatment D) according to the randomization scheme.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment A (Experimental): 600 mg TBPM-PI-HBr (2 x 300 mg tablets) and TBPM-PI-HBr-matching placebo (2 x matching placebo tablets) administered at Hour 0 on Day 1.
  Interventions: Drug: Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) + Placebo; Other: Placebo for Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr)
- Treatment B (Experimental): 1200 mg TBPM-PI-HBr (4 x 300 mg tablets) administered at Hour 0 on Day 1.
  Interventions: Drug: Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr)
- Treatment C (Placebo Comparator): TBPM-PI-HBr-matching placebo (4 x matching placebo tablets) administered at Hour 0 on Day 1.
  Interventions: Other: Placebo for Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr)
- Treatment D (Other): Positive Control - unblinded: 400 mg moxifloxacin (1 x 400 mg tablet) administered at Hour 0 on Day 1.
  Interventions: Drug: Moxifloxacin 400mg

INTERVENTIONS:
Drug: Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) + Placebo — Treatment A: Subjects receive TBPM-PI-HBr + matching Placebo.
  Other Names: SPR994
  Arms: Treatment A
Drug: Moxifloxacin 400mg — Treatment D: Subjects receive 1 400 mg tablet of moxifloxacin administered in an open label manner.
  Other Names: Avelox
  Arms: Treatment D
Other: Placebo for Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) — Treatment C: Subjects receive TBPM-PI-HBr matching placebo.
  Arms: Treatment A; Treatment C
Drug: Tebipenem Pivoxil Hydrobromide (TBPM-PI-HBr) — Treatment B: Subjects receive TBPM-PI-HBr.
  Other Names: SPR994
  Arms: Treatment B

SUMMARY:
This is a randomized, double-blind (with respect to Tebipenem pivoxil hydrobromide [TBPM-PI-HBr]/placebo only), placebo- and active-control, single-dose, 4-way crossover study that will enroll 24 healthy adult male and female subjects. There will be a washout period of at least 7 days between dosing in each period and each subject will receive all 4 treatments over 4 periods in a crossover study design.

DETAILED DESCRIPTION:
This is a randomized, double-blind (with respect to TBPM-PI-HBr / placebo only), placebo- and active-control, single-dose, 4-way crossover study. Twenty-four (24) healthy, adult, male and female subjects will be enrolled. Screening of subjects will occur within 28 days prior to the first dosing.

All subjects will receive a single dose of 4 different study treatments over 4 separate treatment periods, each separated by a 7-day washout period.

On Day 1 of Period 1, subjects will be randomized to 1 of 12 treatment sequences. Sentinel group: In Period 1 only, 4 subjects will be dosed 24 hours prior to the remaining 20 subjects. Each of the 4 subjects from the sentinel group will receive a different treatment.

On Day 1 of each period, subjects will receive a single oral therapeutic dose of TBPM-PI-HBr (Treatment A), supratherapeutic dose of TBPM-PI-HBr (Treatment B), placebo (Treatment C), or moxifloxacin (Treatment D) according to the randomization scheme.

In each period, cardiodynamic ECGs and PK blood samples will be collected pre-dose and for 24 hours post-dose. Safety will be monitored throughout the study by repeated clinical and laboratory evaluations.

Discontinued subjects who have received study drug will not be replaced.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following inclusion criteria to be eligible for participation in the study:

1. Healthy, adult, male or female, 18-65 years of age, inclusive, at screening.
2. Continuous non-smoker who has not used nicotine-containing products for at least 3 months prior to the first dosing and throughout the study, based on subject self- reporting.
3. Body mass index (BMI) ≥ 18.0 and ≤ 32.0 kg/m2 at screening.
4. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or ECGs, as deemed by the PI or designee.
5. No clinically significant history or presence of ECG findings as judged by the PI or qualified designee at screening and prior to dosing of Period 1, including each criterion as listed below:

   1. Normal sinus rhythm (heart rate between 50 and 100 bpm, inclusive);
   2. QTcF interval (Fridericia's correction to the QT interval) ≤ 450 msec;
   3. QRS interval < 110 msec;
   4. PR interval < 220 msec.
6. For a female of childbearing potential: either be sexually inactive (abstinent as a lifestyle) for 3 months prior to the first dosing and throughout the study or be using one of the following acceptable birth control methods:

   * non-hormone releasing intrauterine device for at least 3 months prior to the first dosing and throughout the study.
   * surgical sterilization of the partner (vasectomy for 4 months minimum prior to the first dosing. In addition, female subjects of childbearing potential will be advised to remain sexually inactive or to keep the same birth control method for at least 28 days following the last dose.
7. For a female of non-childbearing potential: must have undergone one of the following sterilization procedures at least 6 months prior to the first dosing:

   * hysteroscopic sterilization (with confirmation of procedure success with hystosalpingogram);
   * bilateral tubal ligation or bilateral salpingectomy;
   * hysterectomy;
   * bilateral oophorectomy;

   or be postmenopausal with amenorrhea for at least 1 year prior to the first dosing and have follicle-stimulating hormone (FSH) serum levels consistent with postmenopausal status.
8. A non-vasectomized, male subject must agree to use a condom with spermicide or abstain from sexual intercourse during the study until 90 days after the last dosing.

   (No restrictions are required for a vasectomized male provided his vasectomy has been performed 4 months or more prior to the first dosing of study drug. A male who has been vasectomized less than 4 months prior to study first dosing must follow the same restrictions as a non-vasectomized male).
9. If male, must agree not to donate sperm from the first dosing until 90 days after the last dosing.
10. Understands the study procedures in the informed consent form (ICF), and be willing and able to comply with the protocol.

Exclusion Criteria:

Subjects must not be enrolled in the study if they meet any of the following criteria:

1. Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of clinically significant medical or psychiatric condition or disease in the opinion of the PI or designee.
3. History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the subject by their participation in the study.
4. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
5. History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s) or related compounds (especially fluoroquinolone-, carbapenem-, penicillin-, and cephalosporin-antibiotics sensitivity).
6. History or presence of any of the following, deemed clinically significant by the PI or designee:

   1. Ventricular pre-excitation syndrome (Wolff-Parkinson White syndrome);
   2. Arrhythmia or history of arrhythmia requiring medical intervention;
   3. Risk factors for Torsade de Pointes (e.g., heart failure, cardiomyopathy, or family history of Long QT Syndrome);
   4. Sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or conduction abnormalities.
7. Allergy to ECG electrode adhesive patches, band aids, adhesive dressing or medical tape.
8. History of epilepsy or seizure disorder.
9. History of known genetic metabolism anomaly associated with carnitine deficiency (e.g., carnitine transporter defect, methylmalonic aciduria, propionic acidemia).
10. Female subjects with a positive pregnancy test or who are lactating.
11. Positive urine drug or alcohol results at screening or first check-in.
12. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
13. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
14. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
15. Estimated creatinine clearance <80 mL/min at screening.
16. Unable to refrain from or anticipates the use of the following drugs beginning 14 days prior to the first dosing and throughout the study:

    * Any drug, including prescription and non-prescription medications , herbal remedies, or vitamin supplements. After first dosing, acetaminophen (up to 2 g per 24 hours) may be administered at the discretion of the PI or designee.
    * Any gastric acid-reducing medications, including but not limited to proton pump inhibitors (e.g., omeprazole, esomeprazole, lansoprazole), histamine-2 receptor antagonists (e.g., nizatidine, famotidine, cimetidine, ranitidine), and antacids (e.g., Alka-Seltzer, Milk of Magnesia, Amphojel, Gelusil, Maalox, Mylanta, Rolaids, Pepto-Bismol).
    * Valproic acid or divalproex sodium.
    * Probenecid.
17. Has been on a diet incompatible with the on-study diet, in the opinion of the PI or designee, within the 30 days prior to the first dosing and throughout the study.
18. Donation of blood or significant blood loss within 56 days prior to the first dosing.
19. Plasma donation within 7 days prior to the first dosing.
20. Participation in another clinical study within 30 days prior to the first dosing. The 30- day window will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of Period 1 of the current study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-19 (Actual); Primary Completion 2020-02-26 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr on the heart rate corrected QT interval (QTc) by assessing concentration-QT (C-QT) relationship using exposure-response modeling. | Pre-dose through 24 hours post-dose
  Holter monitors will be used to collect continuous 12-lead electrocardiogram (ECG) data on Day 1. Triplicate 10-second, 12-lead ECG recordings will be extracted from the Holter monitor data within a 5-minute time window prior to the pharmacokinetic (PK) blood samples collected as close to the exact time point as possible

SECONDARY OUTCOMES:
1. To evaluate the effect of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr on other electrocardiogram (ECG) parameters. | Pre-dose through 24 hours post-dose
  Number of participants with changes in QTc from baseline.
1. To evaluate the effect of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr on other electrocardiogram (ECG) parameters. | Pre-dose through 24 hours post-dose
  Number of participants with changes in QT from baseline.
1. To evaluate the effect of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr on other electrocardiogram (ECG) parameters. | Pre-dose through 24 hours post-dose
  Number of participants with changes in PR interval from baseline.
1. To evaluate the effect of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr on other electrocardiogram (ECG) parameters. | Pre-dose through 24 hours post-dose
  Number of participants with changes in RR interval from baseline.
1. To evaluate the effect of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr on other electrocardiogram (ECG) parameters. | Pre-dose through 24 hours post-dose
  Number of participants with changes in QRS duration from baseline.
1. To evaluate the effect of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr on other electrocardiogram (ECG) parameters. | Pre-dose through 24 hours post-dose
  Number of participants with changes in heart rate (HR) from baseline.
2. To evaluate pharmacokinetics (PK) of tebipenem (TBPM) after administration of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr. | Pre-dose through 24 hours post-dose
  AUC0-last will be calculated for TBPM and moxifloxacin in plasma.
2. To evaluate pharmacokinetics (PK) of tebipenem (TBPM) after administration of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr. | Pre-dose through 24 hours post-dose
  AUC0-inf will be calculated for TBPM and moxifloxacin in plasma.
2. To evaluate pharmacokinetics (PK) of tebipenem (TBPM) after administration of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr. | Pre-dose through 24 hours post-dose
  AUC%extrap will be calculated for TBPM and moxifloxacin in plasma.
2. To evaluate pharmacokinetics (PK) of tebipenem (TBPM) after administration of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr. | Pre-dose through 24 hours post-dose
  Cmax will be calculated for TBPM and moxifloxacin in plasma.
2. To evaluate pharmacokinetics (PK) of tebipenem (TBPM) after administration of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr. | Pre-dose through 24 hours post-dose
  Tmax will be calculated for TBPM and moxifloxacin in plasma.
2. To evaluate pharmacokinetics (PK) of tebipenem (TBPM) after administration of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr. | Pre-dose through 24 hours post-dose
  Kel will be calculated for TBPM and moxifloxacin in plasma.
2. To evaluate pharmacokinetics (PK) of tebipenem (TBPM) after administration of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr. | Pre-dose through 24 hours post-dose
  t1/2 will be calculated for TBPM and moxifloxacin in plasma.
3. To assess the safety and tolerability of a single therapeutic and supratherapeutic dose of TBPM-PI-HBr. | Pre-dose through 24 hours post-dose
  Number of participants with treatment-related adverse events using CTCAE v5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No